CLINICAL TRIAL: NCT01778517
Title: Treatment of Functional Movement Disorders With Psychotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130047; 13-N-0047
Record Dates: First submitted 2013-01-26; First posted 2013-01-29 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2015-07-23

CONDITIONS: Movement Disorders
Keywords: Psychogenic Movement Disorders
MeSH Terms: conditions — Movement Disorders | interventions — Psychotherapy, Group

INTERVENTIONS:
Other: Group Psychotherapy
Other: Cognitive behavior therapy based on self help

SUMMARY:
Background:

- Functional movement disorder (FMD) is a form of conversion disorder (CD). CD is a disorder in which a person has neurological symptoms that do not have a neurological cause. These symptoms can include pain, weakness, dizziness, and fatigue. Some thoughts on CD suggest that it may come from feelings of anxiety that are converted into physical symptoms. Treatment for FMD usually involves stress reduction, family help, and regular doctor s appointments. Therapy interventions, however, have not been well studied. Researchers want to see if people with FMD get better with psychotherapy. They will study two different types of psychotherapy: group therapy and a self-help manual.

Objectives:

- To test two different types of therapy treatments for FMD.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with FMD by a neurologist.

Design:

* Participants will be screened with a physical exam and medical history. They will also have a psychological exam, and answer questions about their mood and symptoms.
* Participants will be separated into three groups. One group will have group therapy. Another will use a self-help workbook designed for people with FMD, and have individual therapy sessions. A third group will just have standard care. During the study, participants will continue to see their regular doctor.
* Group therapy participants will meet once a week for 6 months at the National Institutes of Health clinical center. There will be 8 to 10 people per group. Sessions will last 75 minutes. These sessions will work on methods for treating FMD.
* Self-help workbook participants will have six individual therapy sessions over 3 to 4 months. They will use the workbooks to learn about and practice methods for treating FMD.
* All participants will be evaluated at 3, 6, and 12 months during the study.
* At the end of the study, participants will have a final follow-up session with exams and questions similar to the screening exam. They will return to the care of their regular doctor.

DETAILED DESCRIPTION:
Objectives:

This is an exploratory study of two options for treating functional movement disorders (FMD):

* Group psychotherapy
* Cognitive behavioral therapy (CBT)-based guided self-help.

Study population:

We intend to study adult patients with diagnoses of FMD seen by the Human Motor Control Section Clinic (HMCS) and who live in the Washington-Baltimore metropolitan area for group psychotherapy as well as patients who live out of the area for CBT-based guided self-help.

Design:

Patients will be screened for participation through protocol 07-N-0190 ( Neurobiology of Psychogenic Movement Disorder and Non-Epileptic Seizures ). Those who meet the inclusion criteria and who live locally will be invited to participate in a treatment study of group psychotherapy. The duration of the study for each patient is one year. Local patients who meet the inclusion criteria will be divided into two groups of 10 patients each. Accrual will be gradual. All 10 patients in each group will start simultaneously. All participants will undergo an initial assessment, followed by an assessment at 3, 6, and 12 months. The primary endpoint will be assessed at 6 months. At the end of the study, all subjects will undergo the same MRI studies they completed as part of protocol 07-N-0190 baseline assessment. Patients will be evaluated with the scales described below.

Those who meet the inclusion criteria and who live locally will be invited to participate in a treatment study of group psychotherapy. Local patients who meet the inclusion criteria will be divided into two groups of 10 patients each. Accrual will be gradual. All 10 patients in each group will start simultaneously. All group participants will be asked to sign a therapy contract , a nonbinding group therapy conduct guideline.

Patients who are out-of-town and meet the inclusion/exclusion criteria will be invited to join the CBT-based guided self-help arm. They will be randomized in two groups of 20 patients each. One group will undergo CBT-based guided self-help; the other will be randomized to standard of care. Standard of care is defined as pharmacological or other treatment modalities excluding CBT or group psychotherapy (the studied modalities). Subjects will be included on a rolling basis, and therapy will be delivered approximately once every two weeks for a total of six sessions. Participants will be instructed in the use of CBT-based self-help workbooks aimed at treating functional neurological symptoms (Overcoming unexplained neurological symptoms: a five areas approach by Dr. Chris Williams, 2011, Hodder and Arnold). Total duration of the intervention will be about 6 months. Subjects will undergo the same assessments as patients in the group psychotherapy arm of the study at the same time points. Only participants in the standard of care arm who successfully complete the whole study will be offered the CBT-based guided self-help therapy after study completion.

Outcome measures:

Primary Outcome measure

-Ability to participate in social roles and activities (Neuro-QOL Item Bank) at 6 months after initiation of therapy.

Secondary Outcome Measures

* Clinical global impression of severity (CGI).
* Subjective and objective depressive and anxiety symptoms, measured with the Beck Depression Inventory (BDI), Hamilton Depression Rating Scale-17, State Trait Anxiety Inventory (STAI) and Hamilton Anxiety Scale.
* Patient and physician rated assessment of disease severity (5 point Likert scales).
* Somatic symptoms (SCL-90).
* Insight, measures with the Brown Assessment of Beliefs Scale (BABS)
* Similar measures at 12 months after initiation of therapy.
* MRI studies (resting state BOLD fMRI, DTI, VBM) comparison between baseline (protocol 07-N-0190) and 6 months after initiation of therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must have participated in Protocol 07-N-0190 ( Neurobiological studies of psychogenic movement disorder and non-epileptic seizure )
* Diagnosis of clinically definite FMD utilizing Fahn and Williams criteria. The diagnosis must be made by a neurologist
* Patients who have active movement symptoms at baseline and score at least 20 percent less than the maximum score on the Neuro-QOL Item Bank
* Able to give informed consent
* All participants should be English-speaking
* Age 18 or older
* Willingness to come without reimbursement to treatment visits for up to 6 months
* Willingness to remain on the same medications for the entire duration of the study

EXCLUSION CRITERIA:

* Have significant neurological disorders (primary or comorbid) such as neurodegenerative disorders, stroke, movement disorders or epilepsy
* Patients with psychotic disorders or bipolar disorder
* Patients with history of alcohol and substance use disorders within the last year, as defined by the DSM-IV-TR (nicotine and caffeine use is not criterion for exclusion)
* Current suicidal/homicidal ideation
* Disease severity requiring inpatient treatment. Chronic pain requiring treatment with narcotic medication

ADDITIONAL EXCLUSIONAL CRITERIA FOR MRI:

* Patients with movement symptoms at rest that may substantially inhibit resolution, comfort, or safety of MRI
* Previous history of or MRI findings consistent with brain tumors, strokes, trauma or arterial venous malformations
* History of traumatic brain injury with loss of consciousness or amnesia lasting greater than a few seconds
* Contraindication to MRI
* Pregnancy
* Patients with current post-traumatic stress disorder, panic disorder or obsessive compulsive disorders
* Patients on tricyclic antidepressants or antiepileptic medications.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-12-11; Primary Completion 2015-07-23 (Actual); Study Completion 2015-07-23 (Actual)

PRIMARY OUTCOMES:
Ability to participate in social roles and activities (Neuro-QOL Item Bank) | 6 months

SECONDARY OUTCOMES:
Somatic symptoms (SCL-90). | at baseline
Self assessment of disease severity (5 point Likert scale). | 3 months
Subjective and objective depressive and anxiety symptoms. | 6 months
Clinical Global impression of severity (CGI). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Williams DT, Ford B, Fahn S. Phenomenology and psychopathology related to psychogenic movement disorders. Adv Neurol. 1995;65:231-57. No abstract available. PMID 7872143
- [Background] Carson AJ, Ringbauer B, Stone J, McKenzie L, Warlow C, Sharpe M. Do medically unexplained symptoms matter? A prospective cohort study of 300 new referrals to neurology outpatient clinics. J Neurol Neurosurg Psychiatry. 2000 Feb;68(2):207-10. doi: 10.1136/jnnp.68.2.207. PMID 10644789
- [Background] Feinstein A, Stergiopoulos V, Fine J, Lang AE. Psychiatric outcome in patients with a psychogenic movement disorder: a prospective study. Neuropsychiatry Neuropsychol Behav Neurol. 2001 Jul-Sep;14(3):169-76. PMID 11513100